CLINICAL TRIAL: NCT01380106
Title: A Controlled, Parallel-Group, Randomized, Open-Label Study to Evaluate Two Lenalidomide Dose Regimens When Used in Combination With Low Dose Dexamethasone for the Treatment of Subjects With Relapsed Multiple Myeloma
Brief Title: Study to Evaluate Two Lenalidomide Dose Regimens With Low Dose Dexamethasone for the Treatment Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston VA Research Institute, Inc. (Other)
Collaborators: Celgene Corporation (Industry); Kansas City Veteran Affairs Medical Center (U.S. Federal Agency); VA Pittsburgh Healthcare System (U.S. Federal Agency); VA Greater Los Angeles Healthcare System (U.S. Federal Agency); Michael E. DeBakey VA Medical Center (U.S. Federal Agency); Edward Hines Jr. VA Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nikhil Munshi, M.D., Principal Investigator -- Coordinating site, Boston VA Research Institute, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RV-MM-PI-0345
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Results first posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Relapsed; Revlimid
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lenalidomide 25mg (Active Comparator): Subjects will receive oral lenalidomide 25mg once daily for days 1-21 out of a 28 cycle
  Interventions: Drug: Lenalidomide 25mg
- Lenalidomide 15mg (Active Comparator): Subjects will receive oral lenalidomide 15mg once daily for days 1-21 out of a 28 cycle
  Interventions: Drug: Lenalidomide 15mg

INTERVENTIONS:
Drug: Lenalidomide 15mg — Subjects will receive oral lenalidomide 15 mg once daily for 1-21 of a 28 day cycle.
  Other Names: REVLIMID®
  Arms: Lenalidomide 15mg
Drug: Lenalidomide 25mg — Subjects will receive oral lenalidomide 25mg once daily for days 1-21 out of a 28 cycle
  Other Names: REVLIMID®
  Arms: Lenalidomide 25mg

SUMMARY:
This is a research study to evaluate two different Lenalidomide doses (15 mg vs. 25 mg) in combination with low dose dexamethasone in patients with relapsed multiple myeloma.

The investigators propose to use the need for dose reduction as a criterion to judge tolerability from various causes. In the veteran population which predominantly is in the older age category with number of co-morbidities, a lower dose regimen may be safer and advantageous.

This study expects to enroll approximately 80 subjects from participating VA sites across the nation.

The investigators will evaluate the safety of the two dose regimens by comparing frequency of dose reductions. The investigators will also measure how long the responses last with each dose.

Lenalidomide is approved by the Food and Drug Administration (FDA) for the treatment of specific types of myelodysplastic syndrome (MDS) and in combination with dexamethasone for patients with multiple myeloma (MM) who have received at least 1 prior therapy. MDS and MM are cancers of the blood. It is currently being tested in a variety of cancer conditions. In this case it is considered experimental.

At the time of enrollment, one-half of the subjects will be chosen at random to receive the 15 mg Lenalidomide dose and the other half will take the 25 mg dose regimen of Lenalidomide. Depending on lenalidomide treatment assignment, subjects will receive either 15 mg p.o. q.d. or 25 mg p.o. q.d. for days 1-21 of a 28 day cycle. In addition, dexamethasone (40 mg) will be added once a week (Days 1, 8, 15 and 22) to the Lenalidomide regimen, with a dose reduction on the same schedule if the patient cannot tolerate the higher dose of dexamethasone. ASA (81 or 325mg) will be given daily for anticoagulation prophylaxis. Patients intolerant to ASA may use low molecular weight heparin. Lovenox is recommended. Coumadin will be allowed provided the patient is fully anticoagulate with INR 2.0 to 2.5.

DETAILED DESCRIPTION:
Primary Objective:

• Evaluate the frequency of dose reductions in two different lenalidomide dose regimens.

Secondary Objectives:

* Evaluate the efficacy of two different lenalidomide dose regimens in patients with multiple myeloma using the EBMT and IMWG criteria.
* Evaluate the duration of response of 15 mg Lenalidomide and 25 mg of Lenalidomide when used in combination with Low Dose Dexamethasone.
* Evaluate the safety of 15 mg and 25 mg of Lenalidomide regiments when in combination with dexamethasone.
* Explore blood and cellular levels of angiogenic factors, cytokines, and adhesion molecules.

ELIGIBILITY:
Inclusion Criteria:

1. Previously diagnosed with multiple myeloma.
2. Must have relapsed or refractory disease (refractory is defined as progression during treatment or within 60 days after the completion of treatment) requiring 2nd or 3rd line therapy
3. Patients may have received lenalidomide and/or dexamethasone
4. Patients must have measurable disease:

   * Serum monoclonal protein >0.5g/dL and/or 0.2g/24hr urine light chain excretion
   * Patients with lower M-protein values or non-secretory myeloma will be eligible if measurable disease can be established, such as serum FreeliteTM chain ratio >5x ULN, measurable soft tissue plasmacytoma >2cm by either physical exam and/or applicable radiographs (i.e. MRI, CT-scan) and/or bone marrow involvement >30%
5. Age >=18 years at the time of consent.
6. All necessary baseline studies for determining eligibility must be obtained within 14 days prior to enrollment. Serum pregnancy tests (sensitivity of at least 25 mIU/mL), for females of childbearing potential (WCBP) must be completed. The first test must be performed within 10-14 days, and the second test within 24 hours prior to initiation of lenalidomide.
7. Pre-study ECOG performance status 0-2. Patients with lower performance status based solely on bone pain will be eligible.
8. Adequate liver functions: AST and ALT =< 3xULN, alkaline phosphatase =< 3.0x ULN, except if attributed to tumor, and bilirubin =< 2xULN.
9. Have Amylase =< 2.5x ULN
10. Able to adhere to the study visit schedule and other protocol requirements
11. Must understand and voluntarily sign an informed consent document.
12. Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL 10 - 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree not to father a child and agree to use a condom if his partner is of child bearing potential. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
13. All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®. All counseling will be done through RevAssist®.
14. Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation. Patients intolerant to ASA may use low molecular weight heparin. Lovenox is recommended. Coumadin will be allowed provided the patient is fully anticoagulate with INR 2.0 to 2.5.
15. Patients may receive a bisphosphonate.

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or breast feeding females.(Lactating females must agree not to breast feed while taking lenalidomide).
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Renal insufficiency of creatinine clearance <40mL/min
5. Known hypersensitivity to thalidomide or lenalidomide.
6. Development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
7. Concurrent use of other anti-cancer agents or treatments.
8. Known seropositive for an active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible.
9. Has hemoglobin <8.0g/dL. The use of transfusion with pRBC to correct anemia and meet eligibility criteria will not be allowed.
10. Has an absolute neutrophil count <1.0x10^9/L within 14 days before enrollment
11. Peripheral neuropathy of grade >=3. Patients with painful grade 2 neuropathy are also excluded
12. Has platelet count <75x10^9/L within 14 days before enrollment.
13. Plasma cell leukemia at time of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-08; Primary Completion 2017-09-11 (Actual); Study Completion 2017-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil C Munshi, M.D., Principal Investigator — Boston VA Research Institute, Inc.
Locations (7):
- United States (7):
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - West Los Angeles VA Medical Center, Los Angeles, California
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - VA Boston Healthcare System, Jamaica Plain, Massachusetts
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Pittsburgh VA Medical Center, Pittsburgh, Pennsylvania
  - Houston VA Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lenalidomide 25mg | Lenalidomide 15mg
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 33
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenalidomide 25mg | Lenalidomide 15mg | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 13 | 13 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 16 | 17 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 10 | 11 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 33
M-protein [Mean (Full Range); unit: g/dL] | 3.12 [.47 to 6.9] | 2.74 [0 to 6.9] | 2.93 [0 to 6.9]

OUTCOME MEASURES:

1. Primary Outcome: Serious Adverse Events
Description: Type, frequency, severity and timing of adverse events and their relationship to combination therapy with lenalidomide plus dexamethasone.
  SAE Grade 3 indicates a severe or medically significant but not immediately life threatening; hospitalization or prolongation of hospitalization; disabling; limiting self care ADL SAE Grade 4 indicates a life-threatening consequences; urgent intervention indicated.
  SAE Grade 5 Death related to AE.
Time Frame: Data was collected for each subject for the duration of the participation in the study, ranging between 75 to 475 days.
Population: 33
Measure: Number; unit: Events
Arm/Group | Lenalidomide 25mg | Lenalidomide 15mg
Number analyzed (Participants) | 16 | 17
Events
  SAE Grade 3 | 23 | 23
  SAE Grade 4 | 4 | 1
  SAE Grade 5 | 1 | 0

2. Primary Outcome: Duration Until Best Response (at Least MR or Minimal Response)
Description: Number of days between the first day of the first cycle to best M-protein response, at least Minimal Response or higher (Partial Response, Very Good Partial Response, near Complete Response, Complete Response).
Time Frame: Data was collected for each subject for the duration of the participation in the study, ranging between 75 to 475 days.
Population: 33
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Lenalidomide 25mg | Lenalidomide 15mg
Number analyzed (Participants) | 16 | 17
Days | 280.4 [86.6 to 474.3] | 145.5 [75.7 to 215.3]

ADVERSE EVENTS:
Time Frame: Data was collected for each subject for the duration of the participation in the study, ranging between 75 to 475 days.
Arm/Group | Lenalidomide 25mg | Lenalidomide 15mg
All-Cause Mortality (participants affected / at risk) | 1/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 12/16 | 10/17
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide 25mg (N=16) | Lenalidomide 15mg (N=17)
DVT (Cardiac disorders) | 2 (2) | 2 (2)
Loss of consciousness (General disorders) | 1 (1) | 0 (0)
Hematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Pneumonia (Infections and infestations) | 4 (4) | 3 (3)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Pneumonia
Rectal adenocarcinoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Potassium level change (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Alpha strep infection (Infections and infestations) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypercapnic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Coronary ischemia (Cardiac disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Decreased urination (Endocrine disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Low calcium (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neutropenia (Nervous system disorders) | 1 (1) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
GERD (suspected) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gastric Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Altered mental state (Psychiatric disorders) | 0 (0) | 1 (1)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-02-14): https://cdn.clinicaltrials.gov/large-docs/06/NCT01380106/Prot_SAP_000.pdf